CLINICAL TRIAL: NCT00283426
Title: An Open Clinical Feasibility Study to Evaluate Efficacy and Safety of Soluble Beta-1,3/1,6-Glucan in Thermal Burns
Brief Title: Efficacy and Safety Study of Soluble Beta-1,3/1,6-Glucan in Thermal Burns
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow patient recruitment
Sponsor: Biotec Pharmacon ASA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBG-1-10
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Burns
MeSH Terms: conditions — Burns

INTERVENTIONS:
Drug: Soluble beta-1,3/1,6-glucan

SUMMARY:
The purpose of this study is to determine whether soluble beta-1,3/1,6-glucan is an effective and safe treatment of thermal burns and non-injured skin where skin grafts are harvested.

Hypothesis: Soluble beta-1,3/1,6-glucan will through its immunomodulating activities improve wound healing of thermal burns and non-injured skin where skin grafts are harvested.

DETAILED DESCRIPTION:
In severe cases, burn patients commonly exhibit a clinical picture of systemic inflammation with a variety of manifestations ranging from the presence of tachycardia, tachypnea, fever and leukocytosis, and may progress to refractory hypotension. Shock and multiple organ system dysfunction may subsequently occur. Sepsis, caused by infection or bacteremia, is also a common occurrence and a major complication in burn patients.

After cooling the burned area, pain control is important. Local burn wound care starts with cleansing the wound followed by application of topical agents to prevent infection. Such agents may have adverse local or systemic effects and may impede on the wound healing process itself. The use of synthetic or biologic materials for wound covering is becoming increasingly popular, but most of the clinical information about efficacy of such products are anecdotal.

A primary objective in burn care is to have all wounds healed within 1 month. With longer healing periods, there is an increasing likelihood of developing hypertropic scaring and alterations in pigmentation. The development of an effective wound healing agent would therefore be highly beneficial for the suffering patient in terms of decreased healing time and improved cosmetic results.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* written informed consent

Group A - patients with thermal burns

* partial thickness burns (2nd degree) requiring non-surgical primary treatment
* primarily 5-15% TBSA burns, but burn patients with injury size from 1 to 40% TBSA may be included

or

Group B - patients with thermal burns

* non-grafted partial thickness burns (2nd degree) in patients requiring autotransplantation in the early phase
* primarily 5-15% TBSA burns, but burn patients with injury size from 1 to 40% TBSA may be included

or

Group C - patients with thermal burns

* donor site(s) on the ventral side of the body and limbs in deep partial thickness burns (2nd degree) and/or full thickness burns patients requiring autotransplantation during the first 1-3 weeks after injury
* primarily 5-15% TBSA burns, but burn patients with injury size from 1 to 40% TBSA may be included

Exclusion Criteria:

* inhalation injury to airways and lungs
* chemical or high voltage electrical burn
* pregnancy, lactation
* clinical signs or symptoms of acute infection
* any prescription or non-prescription topical medication administered within one week prior to study start
* hematological and clinical/chemical parameteres judged as unacceptable by the investigator
* donor sites with re-harvesting
* previous treatment with soluble beta-1,3/1,6-glucan
* participation in other clinical studies in the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-01; Study Completion 2007-03

PRIMARY OUTCOMES:
Efficacy parameters:
oedema
bleeding
pain on physical contact
exudation
capillary refill
reepithelialization
rubor
paleness
infectious discharge
smell
adherence of dressing
time since last dressing change
The efficacy parameters will be recorded during regular wound procedures

SECONDARY OUTCOMES:
Safety parameters:
vital signs (heart rate, blood pressure, body temperature)
adverse events
laboratory parameters
The safety parameters will be recorded daily during the first week of treatment and weekly thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Tjostolv Lund, Dr.med., Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway